CLINICAL TRIAL: NCT04486950
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-951 in Healthy Subjects Following Intravenous Administration
Brief Title: A Study of TAK-951 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-951-1004; U1111-1251-9214 (Registry Identifier: WHO)
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteer
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Low Dose): TAK-951 20 mcg Infusion Over 60 Minutes (Experimental): TAK-951 20 microgram (mcg) or TAK-951 placebo-matching, infusion, intravenously, over a period of 60 minutes on Day 1.
  Interventions: Drug: TAK-951; Drug: TAK-951 Placebo
- Cohort 2 (High Dose): TAK-951 1 mg Infusion Over 60 Minutes (Experimental): TAK-951 1 milligram (mg) or TAK-951 placebo-matching, infusion, intravenously, over a period of 60 minutes on Day 1. Dose level will be determined based on safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-951; Drug: TAK-951 Placebo
- Cohort 3: TAK-951 1 mg Infusion Over 120 Minutes (Experimental): TAK-951 1 mg or TAK-951 placebo-matching, infusion, intravenously, over a period of 120 minutes on Day 1. Dose level will be determined based on safety, tolerability and PK data from previous cohorts.
  Interventions: Drug: TAK-951; Drug: TAK-951 Placebo

INTERVENTIONS:
Drug: TAK-951 — TAK-951 intravenous infusion.
Drug: TAK-951 Placebo — TAK-951 placebo-matching intravenous infusion.

SUMMARY:
It is hoped that a medicine called TAK-951 will eventually be used to treat nausea and vomiting. Before then, the sponsor needs to understand how the body processes TAK-951 in healthy adults.

The main aims of this study are as follows:

* To check for side effects from TAK-951 when given at a slow and fast infusion rate.
* To learn how much TAK-951 participants can receive without getting side effects from it.

Participants will receive a single infusion of either TAK-951 or placebo. In this study, a placebo looks like TAK-951 but does not have any medicine in it. Participants will receive either a low dose or high dose of TAK-951. The infusion will take from 1-3 hours.

Participants will stay in the study clinic for about 4 days to receive the study medicine (TAK-951 or placebo) and check for side effects. They will have follow-up visits at the clinic about 2 weeks and 4 weeks after treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-951. The study will evaluate the safety, tolerability and PK of TAK-951 in healthy participants.

The study will enroll approximately 40 healthy participants. Each cohort will have 8 participants to be randomized and a minimum of 3 cohorts will be evaluated. Participants will be randomly assigned (by chance, like flipping a coin) to receive TAK-951 or placebo in a 6:2 ratio in one of the following 3 cohorts, which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Cohort 1 (Low Dose): TAK-951 20 mcg Infusion Over 60 Minutes
* Cohort 2 (High Dose): TAK-951 1 mg Infusion Over 60 Minutes
* Cohort 3: TAK-951 1 mg Infusion over 120 Minutes

Sentinel dosing will be done in first 2 participants in each cohort. The dosing in rest of the cohort will done if there are no significant safety or tolerability concerns. Additional 2 cohorts, each cohort with 8 participants may be added in study to evaluate additional intravenous dosing regimen after clinical data analysis of first 3 cohorts. Dosing of the subsequent cohort will be based on the analysis of the previous cohort's data.

This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 57 days. All participants will return to clinic after 14 and 28 days after the last visit to the clinic for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non-smoker who has not used nicotine- and tobacco-containing products and/or cannabis products for at least 3 months prior to dosing and throughout the study.
2. Body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilogram per square meter (kg/m^2) at screening.
3. Female must be of non-childbearing potential.

Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. Drink alcohol in excess of 21 glasses/units per week for males or 14 glasses/units per week for females, with one unit equal to (=) 150 milliliter (mL) of wine or 360 mL of beer or 45 mL of 45 percent (%) alcohol.
3. Have any tattoos, scars or skin issue at planned IV infusion site which could interfere with dosing.
4. History or presence of:

   * Three (3) or more incidences of vasovagal syncope within the last 5 years prior to screening.
   * Family history of unexplained sudden death or channelopathy.
   * Brugada syndrome (that is, right bundle branch block (RBBB) pattern with ST-elevation in leads V1-V3).
   * Cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction, stroke, sick sinus syndrome, pulmonary congestion, symptomatic or significant cardiac arrhythmia, second-degree AV block type 2, third-degree AV block, prolonged corrected QT interval by Fredericia (QTcF) interval, hypokalemia, hypomagnesemia, or conduction abnormalities;
   * Risk factors for Torsade de Pointes (example, heart failure, cardiomyopathy, or family history of Long QT Syndrome);
   * Any clinically significant ECG findings or medical history including: long or short QT interval with QTcF (over 450 msec or less than 360 msec), bifascicular block or QRS >=120 msec or PR interval greater than (>) 200 msec at screening or Day -1 pre-Hour 0.
   * Documented history of sinoatrial block or sinus pause >=3 seconds.
5. Semi-recumbent blood pressure (average of duplicate) is less than 90/60 millimeter of mercury (mmHg) or greater than 140/90 mmHg at screening.
6. Has an average semi-recumbent heart rate <60 or >100 beats per minute (bpm) (at screening, at Day -1 pre-Hour 0, or at pre-dose Day 1); athletic participants with an average semi-recumbent heart rate <60 bpm can be enrolled only with medical monitor approval. If participant has heart rate <60 bpm Investigator should obtain medical approval from Sponsor.
7. Has orthostatic hypotension defined as a decrease in systolic blood pressure >=20 mmHg or a decrease in diastolic blood pressure >=10 mmHg after 2 minutes of standing when compared with blood pressure from the semi-recumbent position at screening and at Day -1 pre-Hour 0. The semi-recumbent blood pressure will be an average of duplicate measurements.
8. Has postural orthostatic tachycardia, defined as an increase of 30 bpm or heart rate >120 bpm after standing for 2 minutes.
9. Positive urine drug or alcohol results at screening or check-in.
10. Positive urine cotinine at screening or check-in.
11. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
12. Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to dosing and throughout the study. Thyroid hormone replacement medication may be permitted if the participant has been on same stable dose for the last 3 months prior to study drug administration. After dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the Investigator or designee. Hormone replacement therapy will also be allowed.
13. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing and throughout the study.
14. Donation of blood or significant blood loss within 56 days prior to dosing.
15. Plasma donation within 7 days prior to dosing.
16. Has positive results for Coronavirus disease 2019 (COVID-19) testing at screening or check-in.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b603d4db2bf003ab4a3c0

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 07 July 2020 to 27 May 2021.
Pre-assignment Details: Healthy participants were randomized and treated sequentially in Cohorts: 1, 2, 3 and 4 to receive intravenous infusion of TAK-951 20 microgram (mcg), TAK-951 1.0 milligram (mg) or TAK-951 matching placebo (normal saline).
Groups:
- Cohorts 1 to 2, Treatment P1: Placebo Pooled: TAK-951 placebo-matching (0.2 milliliter [ml] normal saline), infusion, intravenously over 60 minutes in fasted condition once on Day 1 in healthy participants.
- Cohort 3, Treatment P2: Placebo: TAK-951 placebo-matching (1 ml normal saline), infusion, intravenously over 120 minutes in fasted condition once on Day 1 in healthy participants.
- Cohort 4, Treatment P3: Placebo: TAK-951 placebo-matching (1 ml normal saline), infusion, intravenously over 180 minutes in fasted condition once on Day 1 in healthy participants.
- Cohort 1, Treatment A: TAK-951 20 mcg: TAK-951 20 mcg, infusion, intravenously over 60 minutes in fasted condition once on Day 1 in healthy participants.
- Cohort 2, Treatment B: TAK-951 1.0 mg: TAK-951 1.0 mg, infusion, intravenously over 60 minutes in fasted condition once on Day 1 in healthy participants.
- Cohort 3, Treatment C: TAK-951 1.0 mg: TAK-951 1.0 mg, infusion, intravenously over 120 minutes in fasted condition once on Day 1 in healthy participants.
- Cohort 4, Treatment D: TAK-951 1.0 mg: TAK-951 1.0 mg, infusion, intravenously over 180 minutes in fasted condition once on Day 1 in healthy participants.
Period: Overall Study
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Started | 4 | 2 | 2 | 6 | 6 | 6 | 6
Completed | 4 | 2 | 2 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who were enrolled and received the full or partial dose of study drug or placebo.
Groups:
- Cohorts 1 to 2, Treatment P1: Placebo Pooled: TAK-951 placebo-matching (0.2 ml normal saline), infusion, intravenously over 60 minutes in fasted condition once on Day 1 in healthy participants.
- Total: Total of all reporting groups
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg | Total
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
  Male | 4 | 2 | 2 | 4 | 6 | 5 | 6 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 4 | 2 | 2 | 6 | 6 | 5 | 4 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 5
  White | 3 | 1 | 2 | 4 | 5 | 4 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 2 | 2 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6
Participants | 1 | 0 | 1 | 3 | 1 | 3 | 1

2. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Sign Values
Time Frame: Baseline up to Day 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12- Lead Electrocardiogram (ECG) Values
Time Frame: Baseline up to Day 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values
Time Frame: Baseline up to Day 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Values
Time Frame: Baseline up to Day 29
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-951
Time Frame: Day 1 pre-dose and at multiple time points (up to 30 hours) post-dose
Population: The pharmacokinetic (PK) analysis set consisted of all participants who received the active study drug and had at least one measurable plasma concentration of TAK-951.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 2.758 (25.1) | 110.4 (11.0) | 127.7 (23.9) | 133.2 (9.5)

7. Secondary Outcome: Ceoi: Plasma Concentration at the End of Infusion for TAK-951
Time Frame: Day 1: at the end of infusion (at 30 hours post-infusion)
Population: The PK analysis set consisted of all participants who received the active study drug and had at least one measurable plasma concentration of TAK-951. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 6 | 6 | 5 | 6
nanogram per milliliter (ng/mL) | 0.5203 (143.2) | 48.95 (15.9) | 37.03 (38.4) | 27.06 (9.1)

8. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-951
Time Frame: Day 1 pre-dose and at multiple time points (up to 30 hours) post-dose
Population: The PK analysis set consisted of all participants who received the active study drug and had at least one measurable plasma concentration of TAK-951.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 2.722 (25.4) | 110.0 (10.8) | 127.2 (24.0) | 132.5 (9.5)

9. Secondary Outcome: T1/2z: Terminal Disposition Phase Half-life for TAK-951
Time Frame: Day 1 pre-dose and at multiple time points (up to 30 hours) post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour | 4.025 (0.7100) | 4.670 (0.5576) | 4.454 (0.5124) | 4.640 (0.3410)

10. Secondary Outcome: λz: Terminal Disposition Phase Rate Constant for TAK-951
Time Frame: Day 1 pre-dose and at multiple time points (up to 30 hours) post-dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: per hour (1/hour)
Arm/Group | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
per hour (1/hour) | 0.1781 (0.040265) | 0.1501 (0.016879) | 0.1574 (0.018543) | 0.1500 (0.010488)

11. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) in Serum
Description: ADA positive was defined as a sample that was evaluated as positive in both the ADA screening and confirmatory assays. ADA positive participants was defined as participants who had at least 1 positive ADA result.
Time Frame: Baseline up to Day 29
Population: The immunogenicity analysis set included those participants from the safety analysis set who had a baseline and at least 1 post-dose immunogenicity sample assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events that started after the first dose of study drug (Baseline) up to Day 29
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Cohorts 1 to 2, Treatment P1: Placebo Pooled | Cohort 3, Treatment P2: Placebo | Cohort 4, Treatment P3: Placebo | Cohort 1, Treatment A: TAK-951 20 mcg | Cohort 2, Treatment B: TAK-951 1.0 mg | Cohort 3, Treatment C: TAK-951 1.0 mg | Cohort 4, Treatment D: TAK-951 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/2 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2 | 1/2 | 3/6 | 1/6 | 3/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1 to 2, Treatment P1: Placebo Pooled (N=4) | Cohort 3, Treatment P2: Placebo (N=2) | Cohort 4, Treatment P3: Placebo (N=2) | Cohort 1, Treatment A: TAK-951 20 mcg (N=6) | Cohort 2, Treatment B: TAK-951 1.0 mg (N=6) | Cohort 3, Treatment C: TAK-951 1.0 mg (N=6) | Cohort 4, Treatment D: TAK-951 1.0 mg (N=6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic heart rate response increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT04486950/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04486950/SAP_001.pdf